CLINICAL TRIAL: NCT06677424
Title: Empirical Distributions of ERP Components Elicited by the NeuroCatch® Platform 2: Development of a Reference Interval Database
Brief Title: NeuroCatch Reference Interval Database
Acronym: RR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthTech Connex Inc. (Industry)
Collaborators: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCI_NCClin_007
Record Dates: First submitted 2024-08-26; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Healthy Controls; Brain Function
Keywords: Brain Scan, NeuroCatch®

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, between-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NeuroCatch® Platform 2 (Other): NeuroCatch® Platform 2 Software enables EEG data collection by recording the data during an audio stimulus presentation (i.e., the NeuroCatch® Scan). The Software plays a 6-min proprietary audio sequence stimulus. The NeuroCatch® software generates unique, randomized audio sequences specifically designed to elicit specific brain responses. Once a NeuroCatch® Scan is complete, the software automatically processes the raw EEG data to generate 6 ERP results and saves the results, the data, and details about the scan to the secure NeuroCatch® server in the cloud.
  While EEG is only collected during the scan, the participant is exposed to the device from the time the cap is placed on the head until it is taken off.
  During the scan, the participant will listen to an auditory stimulus sequence consisting of tones and words. This has been designed and limited to safe audio levels.
  Interventions: Device: NeuroCatch® Platform 2

INTERVENTIONS:
Device: NeuroCatch® Platform 2 — The NeuroCatch® Platform 2, a medical device system developed by NeuroCatch Inc., consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP; brain response to a stimulus) information. The device is approved as a medical device by Health Canada.

SUMMARY:
The purpose of this study is to understand how the brain responds to sounds and words, and how this response varies between individuals. The purpose if this study is to develop data set comparing the results from one individual with those from other members (a reference interval database of NeuroCatch® Platform 2) and to quantify the expected distribution across sex and age. NeuroCatch® Platform 2, is a medical device approved by Health Canada. The plan is to enroll 810 participants, the study includes screening for eligibility and one brain scan. The study is conducted at the Centre for Neurology Studies in Surrey, BC or at its satellite sites ( if required).

DETAILED DESCRIPTION:
Study specific Procedures: Includes a screen for eligibility and a scan visit. The total time 30 minutes to 1 hour for the whole study. The procedures can be completed on the same day or split between two days.

Screening visit (15- 30min, virtual visit): Prior to any procedures being conducted, Informed Consent Form will be reviewed in detail, an opportunity will be given to decide to participate in the study or not and if all the study requirements are met as well as all the questions have been answered, consent form is signed. Participant study eligibility is reviewed including medical history, and brain scan requirements. If participant is eligible, scan visit will be completed. If participant is not eligible no further study procedures will be completed.

Scan visit (15-30 min at the clinic): During the scan visit demographic information ( date of birth, sex, level of education, recent sleep, self-described mood, caffeine intake, alcohol consumption, nicotine usage, psychoactive usage, handedness, first language, profession and current medications) is collected, brain scan safety questionnaire is completed and a brain scan with NeuroCatch® Platform 2 will be completed.

NeuroCatch scan procedure: A cap with the EEG sensors is placed on your scalp and will be adjusted to get good recordings of brain activity. An alcohol pad is used to clean the skin of your forehead, and a plastic syringe tip or wooden dowel to move your hair out of the way to place the EEG sensors/electrodes. A small amount of a conductive gel is applied under each electrode. This takes between 5-20 minutes. Once its all set up, you will be asked to listen to an auditory sequence that is 6 minutes long. During this period, you are asked to sit still and listen to the sounds and the words.

Any information about you obtained from or for this research study will be kept as confidential as possible, All participants will be assigned a participant ID and data will identified using the ID.

ELIGIBILITY:
INCLUSION CRITERIA

1. Any sex, at least 6 years of age or older
2. Able to understand the informed consent/assent form (in English), study procedures and willing to participate in study; participants under 19 must also have a parent/guardian who is able to understand and provide informed consent on their behalf.
3. Able to remain seated and focused for 7 minutes
4. In good health with no history of clinically relevant neurological illness or injury

EXCLUSION CRITERIA

1. Requires the use of hearing aids or a cochlear implant, diagnosed with tinnitus that is currently active, or has temporary damage to hearing (e.g., punctured ear drum). Or unable to detect a 740Hz tone played at 85dB in both ears.
2. Implanted pacemaker or other electrical stimulator(s)
3. Metal or plastic implants in the skull, excluding dental/facial implants.
4. Not native-level in English
5. Previous exposure to the NeuroCatch® Platform 2 audio sequences in the last 3 months
6. History of clinically relevant neurological disorders or injury (e.g., epilepsy, Parkinson's disease, traumatic brain injury, etc.)
7. History of chronic pain or chronic headache disorders (e.g. migraine, tension headaches, fibromyalgia, etc.)
8. Currently diagnosed with any sleeping disorders (e.g. sleep apnea, hypersomnia, insomnia, parasomnia, etc.)
9. Diagnosed with any memory disorders.
10. History of clinically relevant major psychiatric disorders (e.g., schizophrenia, bipolar disorder, etc.)
11. History of alcohol or substance misuse that, in the opinion of the Investigator, may impact brain function
12. Use of medications that affect brain function (e.g., antiepileptic drugs, antipsychotics, stimulants, etc.)
13. Serious medical conditions affecting brain functions (e.g., stroke, brain tumor, neurodegenerative diseases, etc.)
14. Undergoing chemotherapy or any form of intensive long-term therapy that, in the opinion of the Investigator, may impact brain function.
15. Unhealthy scalp (e.g., apparent open wounds and/or bruised or weakened skin)
16. Allergy to EEG gel

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Amplitude & Latency collection for NeuroCatch® Platform 2 | 20 minutes
  Response size (amplitude in microvolts) and response timing (latency in milliseconds) will be collected for the ERPs N100, P300 and N400.
Demographic indicators | 5 minutes
  Demographic indicators to be collected such as year of birth, sex, level of education.

SECONDARY OUTCOMES:
Assessing Influences on Brain Function: NeuroCatch® to Lifestyle and Health Factors | 5 minutes
  Measurements include: current medications, mood, total sleep hours, caffeine and alcohol intake, nicotine and psychoactive substance use, as well as any medications taken within 24 hours before the scan, noting whether each is more, less, or equal to the participant's typical amount.

OTHER OUTCOMES:
Safety assessments | 30 minutes
  Safety assessments will me assessed by subjective report of incidence and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Venter, MD, Principal Investigator — Centre for Neurology Studies
Locations (1):
- Centre for Neurology Studies, 13761 96 Ave, Unit 1004, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The study is live, if you are interested learning or want to participate to sign up via the URL hereto let us know you are interested. — https://centreforneurologystudies.com/neurocatch-reference-range-study/